CLINICAL TRIAL: NCT05354765
Title: Exploration of Adaptive Antitumoral Immune Cells Through Lymphapheresis in Cancer Patients : ALCYTA
Acronym: ALCYTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: IC 2020-12
Record Dates: First submitted 2022-04-20; First posted 2022-04-29 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Immune System or Toxicities Suspected
Keywords: tumor-antigen specific immune cells; circulating tumor DNA
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first type, called "A" Cohorts (Experimental): The first type, called "A" Cohorts, corresponds to indications for which the treatment induces a high response rate (>30%). These patients will have a lymphapheresis before and during treatment with immunotherapy. In addition, a blood sample in CellSave® tubes (15mL) will be taken at baseline and three weeks, and EDTA tubes (15mL) will be taken at baseline, 3 weeks after treatment start and at progression.
  Interventions: Other: blood sample
- second type, called "B" Cohorts (Experimental): The second type, called "B" Cohorts, corresponds to indications for which a role of the immune system is suspected. Only the so-called "informative" patients (responders or surprising evolution) will have one lymphapheresis during treatment. The lymphapheresis will be performed between 8 weeks and 18 months after the start of treatment and depending on the clinical course determined by the clinicians in consultation with at least one immunologist (Olivier Lantz, Emanuela Romano, Cécile Alanio, Marion Alcantara).
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — lymphapheresis before and during treatment, blood sample in CellSave® tubes (15mL) will be taken at baseline and three weeks, and EDTA tubes (15mL) will be taken at baseline, 3 weeks after treatment start and at progression
  Arms: first type, called "A" Cohorts
Other: blood sample — lymphapheresis will be performed between 8 weeks and 18 months after the start of treatment
  Arms: second type, called "B" Cohorts

SUMMARY:
The study will evaluate the detection of tumor-antigen specific immune cells in cancer patients in whom the role of the immune system is suspected.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 or over,
2. Patient presenting an invasive tumor pathology (proven or suspected). The location and / or stage of which are defined for each cohort through an amendment to the protocol,
3. Patient treated with immune-modulators or other treatments likely to modify immunological parameters,
4. Suspicion of immune mediated response or toxicities (assessed by the immunologists),
5. Peripheral venous capital usable and compatible with the realization of 2 venous accesses for lymphapheresis and absence of cardiovascular problem (heart failure, arrhythmia ...), per investigator assessement,
6. Total circulating lymphocytes> 1000 / mm3,
7. Availability of DNA and RNA from the tumor,
8. Information to the patient and signature of informed consent or his legal representative,
9. Affiliated with a social security scheme or such a scheme.

Exclusion Criteria:

1. Inability to undergo study follow-up for geographical, social or psychological reasons,
2. Infection with HIV or hepatitis B or C viruses,
3. Patients on high dose corticosteroid treatment (> 1 mg / kg continuously),
4. Any concomitant serious illness that may interfere with participation in the study or significantly affect the results of the study (pulmonary, heart or liver disease),
5. Contraindication to performing lymphapheresis (coagulation disorder, cardiovascular problems, venous access, hypocalcemia, psychological inability to undergo extracorporeal circulation, cachexia, etc.),
6. Pregnant patient or of childbearing age without effective contraception,
7. Persons deprived of their liberty, under guardianship or legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2026-09-03 (Estimated); Study Completion 2026-09-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the presence of tumor-antigen specific T cells for Cohorts A | before treatment
  Presence of tumor-antigen specific T cells using multiplex tetramers and ELISPOTs.
Evaluation of the presence of tumor-antigen specific T cells for Cohorts A | During treatment
  Presence of tumor-antigen specific T cells using multiplex tetramers and ELISPOTs.
Evaluation of the presence of tumor-antigen specific T cells for Cohorts A | at baseline
  Presence of tumor-antigen specific T cells using multiplex tetramers and ELISPOTs.
Evaluation of the presence of tumor-antigen specific T cells for Cohorts A | 3 weeks after treatment start
  Presence of tumor-antigen specific T cells using multiplex tetramers and ELISPOTs.
Evaluation of the presence of tumor-antigen specific T cells for Cohorts A | at progression (up to 100 weeks)
  Presence of tumor-antigen specific T cells using multiplex tetramers and ELISPOTs.
Evaluation of the presence of tumor-antigen specific T cells for Cohorts B | between 8 weeks and 18 months after the start of treatment
  Presence of tumor-antigen specific T cells using multiplex tetramers and ELISPOTs.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Curie, Paris
  - Institut Curie, Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).